CLINICAL TRIAL: NCT03678337
Title: Prevention and Pharmacological Management of Cardiac Adverse Drug Reactions Induced by Drugs Used in Oncology. The PICARO Cohort
Brief Title: Prevention and Pharmacological Management of Cardiac Adverse Drug Reactions Induced by Drugs Used in Oncology.
Acronym: PICARO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00429-46
Record Dates: First submitted 2018-08-13; First posted 2018-09-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-08

CONDITIONS: Cardio-oncology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort with plasma samples
  Interventions: Other: observational cohort with plasma samples

INTERVENTIONS:
Other: observational cohort with plasma samples — plasma samples

SUMMARY:
Recently, the medical management of cancer patients has considerably improved the prognosis of these patients and today some cancers are becoming "chronic diseases". As a result, new adverse effects (AEs) are observed, particularly cardiac.

These "new" cardiac AEs are the consequence of a significant increase in patients life expectancy (delayed AEs not previously seen) but also the use of new pharmacological classes of anticancer drugs such as kinase inhibitors. The incidence of these cardiac AEs varies according to the patient profile and the anticancer molecules used, but their impact on the morbidity and mortality of the patients is significant.

In this context, we started at the University Hospital of Caen Normandy in September 2017 a cardio-oncology program entitled "prevention and pharmacological management of cardiac adverse effects induced by drugs used in Oncology" (PICARO program). This program involves the pharmacology department (opening of a dedicated consultation), the cardiology department (opening of a dedicated ultrasound consultation), vascular medicine departement (opening of a dedicated consultation) and the oncology federation. This program aims to be regional in the future. We therefore propose to build a cohort backed up to the PICARO program to assess the regional impact of cardiac AEs of anticancer drugs and thus to be better able to specify the number of AEs, the incidence and regional prevalence of these drugs. .

The constitution of this cohort is only the first step towards the constitution in the near future (2 years) of an observatory and then a regional registry of cardiac AEs induced by anticancer drugs. The objectives associated with the establishment of such a registry would be to reduce the number of cardiac AEs, the hospitalizations caused by these AEs, a better information of health professionals and patients, an improvement in the screening of patients at risk, all coming back in the context of health, clinical, epidemiological and pharmacological surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years,
* Attents of cancer,
* Addressed for the first time to one of the PICARO program consultations at the University Hospital of Caen Normandy,
* Written informed consent,
* Patient beneficiary of the french social insurance.

Exclusion Criteria:

* Minor and major protected patients
* pregnant or nursing women
* patient already included in the PICARO cohort
* Patients under guardianship, curatorship, safeguard of justice or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cancer patients presenting the eligibility criteria referred to the PICARO program
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-09-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With AntiCancer Drugs-Related Cardiac Adverse Events during the follow-up | 2 years

SECONDARY OUTCOMES:
Plasmatic tests to predict anticancer drugs-related cardiac adverse events from the constitution of the plasma biobank | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolladille C, Ederhy S, Allouche S, Dupas Q, Gervais R, Madelaine J, Sassier M, Plane AF, Comoz F, Cohen AA, Thuny FR, Cautela J, Alexandre J. Late cardiac adverse events in patients with cancer treated with immune checkpoint inhibitors. J Immunother Cancer. 2020 Jan;8(1):e000261. doi: 10.1136/jitc-2019-000261. PMID 31988143